CLINICAL TRIAL: NCT03147404
Title: SAMSUND MEDICAL CENTER
Brief Title: Phase II Study of Avelumab in Metastatic Gastronetro-pancreatic （GEP） Neuroendocrine Carcinoma （NEC, WHO Grade 3） as Second-line Treatment After Failing to Etoposide+Cisplatin: Integration of Genomic Analysis to Identify Predictive Molecular Subtypes
Acronym: MS100070-0177
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Seung tae Kim, Samsung Medical Center, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-04-085
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Neuroendocrine Carcinoma, Grade 3
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Lymphoma, Follicular | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: Avelumab 10 mg/kg i.v. every 2 weeks (Q2W)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab 10 mg/kg i.v. every 2 weeks (Q2W)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/kg i.v. every 2 weeks (Q2W)
  Other Names: Bavencio

SUMMARY:
Phase II study of avelumab in metastatic gastronetro-pancreatic (GEP) neuroendocrine carcinoma (NEC, WHO grade 3) as second-line treatment after failing to etoposide+cisplatin: integration of genomic analysis to identify predictive molecular subtypes

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of up to 28 days, eligible subjects will receive treatment beginning on Day 1 of each 2-week dosing cycle for aveluumab. Treatment with aveluumab will continue until documented disease progression, unacceptable adverse event(s),intercurrent illness that prevents further administration of treatment, Investigator's decision to withdraw the subject, subject withdraws consent, pregnancy of the subject, noncompliance with trial treatment or procedure requirements, After the end of treatment, each subject will be followed for 30 days for adverse event monitoring (serious adverse events and events of clinical interest will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier). Subjects who discontinue after 24months of therapy for reasons other than disease progression or intolerability or who discontinue after attaining a CR may be eligible for up to one year of retreatment after they have experienced radiographic disease progression. Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up for disease status until disease progression, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival until death, withdrawal of consent, or the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial. The subject may also provide consent for Biomedical Research. However, the subject may participate in the main trial without participating in Biomedical Research.
2. Be20 years of age on day of signing informed consent
3. Have histologically or cytologically-confirmed diagnosis of GEP-NECs including all gastrointestinal tracts
4. Have metastatic disease or locally advanced, unresectable disease with feasible biopsy sites (baseline and follow up)
5. Has experienced documented objective radiographic or clinical disease progression during or after first-line therapy containing any platinum/etoposide
6. Have measurable disease based on mRECIST as determined by investigator. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has grade 1 or 2 neuroendocrine tumor in GI tracts.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active TB
5. Hypersensitivity to avelumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
BEST OF RESPONSE | 12months

SECONDARY OUTCOMES:
OVERALL RESPONSE | 24months

CONTACTS AND LOCATIONS:
Overall Officials: SeungTae KIM, MD, Ph.D, Principal Investigator — SamsungMedicalCenter
Locations (1):
- Samsung Medical Center, Seoul, South Korea